CLINICAL TRIAL: NCT00438360
Title: A 24-week, Double-blind, Randomized, Placebo-controlled, Multicenter Study, to Evaluate the Effectiveness of Cyclosporine 2,5 mg/kg/Day Bid Twice a Week on Reducing Relapse Rate, in Maintenance Patients With Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Cyclosporine A Microemulsion in Maintenance Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLO400CIT04
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Cyclosporine, chronic plaque psoriasis, intermittent therapy
MeSH Terms: interventions — Cyclosporine

ARMS (2):
- Cyclosporine A (Active Comparator): Oral soft gelatin capsules of cyclosporine 10 mg, 25 mg, 50 mg or 100 mg administered twice a week for 24 weeks at the dosage of 5 mg/Kg/day in two daily administrations
  Interventions: Drug: Cyclosporine A microemulsion
- Placebo (Placebo Comparator): Oral soft gelatin capsules of placebo matching cyclosporine administered twice a week for 24 weeks in two daily administrations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine A microemulsion — Oral soft gelatin capsules of Cyclosporine 10 mg, 25 mg, 50 mg or 100 mg administered twice a week for 24 weeks at the dosage of 5 mg/Kg/day in two daily administrations
  Other Names: Neoral
  Arms: Cyclosporine A
Drug: Placebo — Oral soft gelatin capsules of placebo matching cyclosporine administered twice a week for 24 weeks in two daily administrations
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of cyclosporine at 2, 5 mg/kg/day bid (i.e. bis in a day), when administered twice a week compared to continuous administration, in patients with chronic plaque psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Outpatients 18 years of age and older (max 65 years)
* Patients with chronic plaque psoriasis on disease remission (i.e. PASI ≤75% of PASI before cyclosporine continuous treatment course) entering a maintenance period
* Disease remission obtained with only cyclosporine as systemic therapy (maximum dose 5 mg/kg/day) for >8 weeks and <16 weeks
* PASI still <75% of PASI before cyclosporine continuous treatment course, at randomization to study treatment (8±2 days after disease remission)

Exclusion criteria:

* Abnormal renal function (creatinine ≥ 10% the upper limit of the reference range)
* Severe chronic degenerative diseases
* Severe uncontrolled hypertension
* Body weigh >110 kg
* Abnormal liver function
* Hyperkalemia or hyperuricemia
* Clinically significant impairment of hematopoietic and cardiovascular function
* Concomitant therapy with nephrotoxic medications
* Patients with malignancy or a history of malignancy
* Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception
* Clinically significant uncontrolled bacterial, viral or fungal infection
* Evidence of drug and/or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Bari, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclosporine A | Placebo
Started | 162 ("Started" indicates randomized patients.) | 81
Intention to Treat (ITT) Population | 160 (These numbers are different from those started (randomized) as 2 pts from each arm never took drug.) | 79
Completed | 90 | 38
Not Completed | 72 | 43
Not completed — Adverse Event | 6 | 1
Not completed — Lack of Efficacy | 42 | 27
Not completed — Other | 24 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine A | Placebo | Total
Number analyzed (Participants) | 160 | 79 | 239
Age, Customized [Number; unit: Participants] — Baseline measures are based on intention to treat (ITT) population.
  Participants
    between 18-45 years | 100 | 48 | 148
    Between 46 and 65 years | 59 | 29 | 88
    >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 32 | 87
  Male | 105 | 47 | 152

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse Rate (Success or Failure), as Assessed by Psoriasis Area and Severity Index (PASI) Score
Description: PASI is an index used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of severest degree. Relapse is considered a worsening of psoriasis associated to a PASI score >75% of PASI score recorded before starting induction therapy with CsA (before study start). Each patient was considered as failure (relapse occurrence) if rate was >= 75%. In all the other cases the patient was considered as success (no relapse).
Time Frame: 24 weeks
Population: Intent to treat population.
Measure: Number; unit: Participants
Arm/Group | Cyclosporine A | Placebo
Number analyzed (Participants) | 160 | 79
Participants
  Success at 6 months | 87 | 36
  Failure at 6 months | 73 | 43

2. Secondary Outcome: Proportion of Participants With Clinical Relapse
Description: Clinical relapse was defined as worsening of psoriasis associated with a Psoriasis Area and Severity Index (PASI) >75% of the PASI score assessed before the continuous treatment, or when the investigator or the patient judged it necessary to change the treatment.
Time Frame: 24 weeks
Population: Intent to treat population.
Measure: Number; unit: proportion of participants
Arm/Group | Cyclosporine A | Placebo
Number analyzed (Participants) | 160 | 79
proportion of participants | 0.369 | 0.456

3. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: PASI is an index used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (best) to 72 (worst), with the highest score representing complete erythroderma of the severest degree.
Time Frame: baseline and week 24
Population: Intention to treat (ITT) population. Patients with a value of PASI at baseline and 24 weeks were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cyclosporine A | Placebo
Number analyzed (Participants) | 158 | 76
Units on a scale | 5.70 (8.0) | 6.86 (8.4)

4. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis
Description: BSA is a measure of the percentage of body surface affected by psoriasis. Using the Mosteller Formula: BSA = BSA (m²) = ( [Height(in) x Weight(lbs) ]/ 3131 )½ . A covariance analysis was performed on all variables, with value assessed at visit 2 as covariate and center as effect. For each variable the changes versus the last available measures were computed
Time Frame: Baseline and week 24
Population: Intent to Treat (ITT) population. Patients with a value of BSA at baseline and 24 weeks were included in this analysis.
Measure: Mean (Standard Deviation); unit: BSA (m^2)
Arm/Group | Cyclosporine A | Placebo
Number analyzed (Participants) | 158 | 76
BSA (m^2) | 8.12 (12.9) | 10.45 (16.7)

5. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Patient Self Assessment of Pruritus
Description: Target lesion pruritus as measured by the Visual Analog Scale (VAS) from 0 to 100 mm at week 24 compared to baseline (with 0 being no pruritis and 100 being maximum pruritis).
Time Frame: Baseline and week 24
Population: Intent to treat (ITT) population. Patients with a value of VAS at baseline and 24 weeks were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cyclosporine A | Placebo
Number analyzed (Participants) | 158 | 76
Units on a scale | 17.32 (30.9) | 25.44 (31.9)

6. Secondary Outcome: Safety / Tolerability Assessed by Adverse Events
Time Frame: 24weeks
Reporting Status: Not Posted
Measure: Number; unit: patient

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Safety Population
Arm/Group | Cyclosporine A | Placebo
Serious Adverse Events (participants affected / at risk) | 1/160 | 0/79
Other Adverse Events (participants affected / at risk) | 19/160 | 1/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine A (N=160) | Placebo (N=79)
Breast mass (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine A (N=160) | Placebo (N=79)
Abdominal pain upper (Gastrointestinal disorders) | 12 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.